CLINICAL TRIAL: NCT03733002
Title: Efficacy and Safety of AngongNiuhuang Pill for the Treatment of Patients With Acute Ischemic Stroke.
Acronym: AGNH2018
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: China-Japan Friendship Hospital (Other); Cangzhou Central Hospital (Other); The Second Hospital of Hebei Medical University (Other); Affiliated Hospital of Chengde Medical University (Other)
Responsible Party: Principal Investigator, Bin Peng, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PUMCH-AGNH2018
Record Dates: First submitted 2018-11-01; First posted 2018-11-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; AngongNiuhuang pill
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AngongNiuhuang (Experimental): Drugs: AngongNiuhuang pill. The other treatments will be provided according to guidelines for standard treatment of acute ischemic stroke.
  Interventions: Drug: AngongNiuhuang pill; Other: Standard treatment
- Placebo of AngongNiuhuang (Placebo Comparator): Drugs: Placebo of AngongNiuhuang pill. The other treatments will be provided according to guidelines for standard treatment of acute ischemic stroke.
  Interventions: Drug: Placebo of AngongNiuhuang pill; Other: Standard treatment

INTERVENTIONS:
Drug: AngongNiuhuang pill — This group will receive AngongNiuhuang pill 1 pill 1 times/day for 5-day.
  Arms: AngongNiuhuang
Drug: Placebo of AngongNiuhuang pill — This group will receive Placebo of AngongNiuhuang pill 1 pill 1 times/day for 5-day.
  Arms: Placebo of AngongNiuhuang
Other: Standard treatment — The other treatments according to guidelines for standard treatment of acute ischemic stroke.

SUMMARY:
AngongNiuhuang pill has obvious effects on the cardiovascular and cerebrovascular, especially the cerebral vessels. Pharmacological experiments confirmed that AngongNiuhuang pill can protect blood-brain barrier, reduce capillary permeability, improve the tolerance of cerebral ischemia and hypoxia, improve oxidative stress injury, thus protecting brain tissue. Clinical studies have also confirmed that AngongNiuhuang pill can increase the GCS score, reduce coma, improve nerve function defect and promote nerve function recovery. The primary purpose of this trial was to evaluate the effect of AngongNiuhuang pill and placebo on the improvement of life function in patients with ischemic stroke at 90 days in acute phase.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, double-blinded, placebo parallel controlled, multiple-center trial. A total of approximately 100 patients (18 years ≤age ≤80 years) within 24 hours of symptom onset of acute ischemic stroke, who shows NIHSS from 5-20 points. Patients fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomized 1:1 into two groups after offering informed content: 1) one group will receive AngongNiuhuang pill 1 pill 1 times/day for 5-day; 2) the other group will receive Placebo of AngongNiuhuang pill 1 pill 1 times/day for 5-day.The primary purpose of this trial was to evaluate the effect of AngongNiuhuang pill and placebo on the improvement of life function in patients with ischemic stroke at 90 days in acute phase. The study consists of five visits including the day of randomization, 2-6 days, monitor daily temperature, 7 days when the therapy is done, 30 days, and 90 days when the follow-up is finished. Demographic information, symptoms and signs, laboratory test, neuro-imaging assessment neurological function rating scale will be recorded during the program. The improvement of life function will be assessed by Modified Rankin Scale(namely score=0-2). The trial is anticipated to last from July 2018 to December 2019 with 100 subjects recruited form 5 centers in China. All the related investigative organization and individuals will obey the Declaration of Helsinki and Chinese GCP standard. A Data and Safety Monitoring Board (DSMB) will regularly monitor safety during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke.
2. 18 years ≤ age ≤ 80 years.
3. Within 24 hours from symptom onset.
4. Baseline NIHSS range 5 from 20.
5. Provision of informed consent.

Exclusion Criteria:

1. Not suitable for taking this medicine after dialectic of traditional Chinese medical doctor.
2. Suffering from intracranial tumors, encephalitis, subarachnoid hemorrhage and other brain organic diseases.
3. Receive thrombolysis or endovascular treatment.
4. mRS>1 at randomization (pre-morbid historical assessment).
5. Thrombocytopenia(<100×10*9/L) , hematologic diseases and other systemic bleeding tendency.
6. Sleepy head (GCS≤7).
7. Alanine transaminase > 1.5 times normal upper limit or Aspartate aminotransferase > 1.5 times normal upper limit.
8. Glomerular filtration rate<60 ml/min/1.73m2.
9. Patients who have been taking AngongNiuhuang pills within 3 months.
10. Pregnancy or lactation, women in childbearing age with negative pregnancy test refuse to accept contraception.
11. Participate in clinical studies of other research drugs within the last 30 days.
12. Patients with a life expectancy of less than three months.
13. Incapable to follow this study for mental illness, cognitive or emotional disorders.
14. Unsuitable for this study in the opinion of the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieve favorable clinical outcomes assessed by Modified Rankin Scale(namely score=0-2) | 90days
  Modified Rankin Scale score changes (continuous) and dichotomized at percentage with score 0-2 vs. 3-6 at the 90 days follow-up.
Severity Adverse Event | 90days
  The percentage of the Severity Adverse Events within the 90 days of the therapy.

SECONDARY OUTCOMES:
The proportion of patients achieve favorable clinical outcomes assessed by Modified Rankin Scale(namely score=0-2) | 7days, 30days
  Modified Rankin Scale score changes (continuous) and dichotomized at percentage.
Neurological recovery | 7 days, 30 days,90 days
  The recovery of neurological deficits assessed by the change of the 7days, 30 days and the 90 days NIHSS to the baseline NIHSS.
Barthel Index | 30 days, 90 days
  Change in the score of the Barthel Index.（The Barthel Index (BI) measures 10 basic aspects of self-care and physical dependency, including 10 subscales: feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers, mobility, and stairs. Every subscale ranges from 0 to 10. Its total score range is 0-100. A normal score is 100, and lower scores indicate increasing disability.）
Recurrent stroke, death and other vascular events | 30 days, 90 days
  The quantity of patients who has recurrent stroke, death and other vascular events.
Changes of biomarker (hs-CRP) | 7 days
  Evaluation of the change in (centralization blood sample determination).
Changes of biomarker (IL-10) | 7days
  Evaluation of the change in IL-10 (centralization blood sample determination).
Changes of biomarker (TNF-α) | 7days
  Evaluation of the change in TNF-α level (centralization blood sample determination).
Adverse Events | 7 days, 90 days
  The percentage of the Adverse Events during the therapy.
Severity Adverse Event | 7days
  The percentage of the Severity Adverse Events during the therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Peng, MD, Principal Investigator — Peking Union Medical College
Locations (1):
- Bin Peng, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No